CLINICAL TRIAL: NCT05855057
Title: A Retrospective Single Centered Cohort Study Comparing The Effectiveness of Ultrasound-Guided PCNL Different Positions in Renal Stones Treatment
Brief Title: Effectiveness of US-Guided PCNL Different Positions in Renal Stones Treatment
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abou Elezz Abdel Fattah, Lecturer of Urology, Faculty of Medicine, Benha University, Benha, Egypt, Benha University
Other Study IDs: RC 14-4-2023
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Percutaneous Nephrolithotomy; Renal Stones; Ultrasound Therapy; Complications
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Flank suspended supine position percutaneous nephrolithotomy: This group included 41 patients in flank suspended supine position percutaneous nephrolithotomy.
  Interventions: Procedure: Flank suspended supine position percutaneous nephrolithotomy
- Supine percutaneous nephrolithotomy group: This group included 41 patients in supine percutaneous nephrolithotomy.
  Interventions: Procedure: Supine percutaneous nephrolithotomy group
- Prone percutaneous nephrolithotomy group: This group included 41 patients in prone percutaneous nephrolithotomy.
  Interventions: Procedure: Prone percutaneous nephrolithotomy group

INTERVENTIONS:
Procedure: Flank suspended supine position percutaneous nephrolithotomy — The patients will be placed in the supine position with the shoulder and the buttock will be raised by a 3-l bag of water suspending the flank of the affected side. The body contour will be aligned to the edge of the table. The operating table will be adjusted to the jack knife position, with the tip of the lower part of the table will be slightly lowered. The leg of the affected side of the patent will be straightened dorsally flexed and slightly inner rotated, with the knee of the other side will be flexed. The patients will be then immobilized at the chest and the pelvis with two adherent tapes which crossed each other at the abdomen to form a 'V' shape.
  Groups: Flank suspended supine position percutaneous nephrolithotomy
Procedure: Supine percutaneous nephrolithotomy group — The patient will remain in the supine position, with the side of interest at the edge of the table, with a small cushion placed under the flank to elevate it 15-20°.
  Groups: Supine percutaneous nephrolithotomy group
Procedure: Prone percutaneous nephrolithotomy group — Prone percutaneous nephrolithotomy. The prone position (PRON) technique followed these classic steps: patients will be placed in a lithotomy position and a ureteral catheter will be inserted through a rigid cystoscope to perform a retrograde pyelogram. The ureteral catheter will be fixed to a Foley catheter, and then the patient will be repositioned to the prone position with pads under their shoulders.
  Groups: Prone percutaneous nephrolithotomy group

SUMMARY:
The aim of this study is to compare the effectiveness of Ultrasound-Guided Percutaneous nephrolithotomyin different positions supine, prone positions and flank suspend supine position in renal stones treatment.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) has become the choice of modality for the treatment of large and complicated renal calculi. Initially, percutaneous access to the kidney was only performed in the prone position, as described sixty years ago.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent Percutaneous nephrolithotomy
* Patient's age from >18 - 70 years old.
* Body mass index (30-40 kg/m2).
* Both sex
* Renal stones diameter ≥2 cm
* Cardiac patients

Exclusion Criteria:

* Patient refusal.
* Pregnant women.
* Patients with renal anomalies.
* Transplanted kidney.
* Uncorrected coagulopathy, or active infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 123 patients who underwent Percutaneous nephrolithotomy at the period from 2018 to 2022 and were diagnosed with consecutive, adult obese patients (age >18-70 years) with renal stones diameter ≥2 cm
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Stone clearance rate | 3 months postoperatively
  Comparison of stone clearance rates among different positions (flank suspended supine, supine, and prone) in Ultrasound-Guided Percutaneous Nephrolithotomy (PCNL) for the treatment of renal stones.

SECONDARY OUTCOMES:
Operative time | Intraoperatively
  duration of the Ultrasound-Guided Percutaneous Nephrolithotomy (PCNL) procedure among different positions
Complication rates | 48 hours Postoperatively
  Comparison of postoperative complications (e.g., bleeding, infection, injury) among the different positions.
Stone-free rates | 48 hours Postoperatively
  Comparison of the percentage of patients achieving complete stone clearance among the different positions.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospitals, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study will be available under a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the end of the study.